CLINICAL TRIAL: NCT04232969
Title: A Randomised, Double Blind, Parallel Group, Placebo Controlled, Phase 3 Trial of Exenatide Once Weekly Over 2 Years as a Potential Disease Modifying Treatment for Parkinson's Disease
Brief Title: Exenatide Once Weekly Over 2 Years as a Potential Disease Modifying Treatment for Parkinson's Disease
Acronym: Exenatide-PD3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/0320
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Exenatide; Parkinson's research
MeSH Terms: conditions — Parkinson Disease | interventions — Exenatide

STUDY DESIGN:
Intervention Model Description: A randomised, double blind, parallel group, placebo controlled, Phase 3 trial of Exenatide once weekly over 2 years as a potential disease modifying treatment for Parkinson's disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exenatide (Active Comparator): Exenatide extended release 2mg (Bydureon) once weekly for 96 weeks n=100
  Interventions: Drug: Exenatide extended release 2mg (Bydureon)
- Placebo (Placebo Comparator): Exenatide extended release placebo once weekly for 96 weeks n=100
  Interventions: Drug: Exenatide extended release 2mg (Bydureon)

INTERVENTIONS:
Drug: Exenatide extended release 2mg (Bydureon) — Subcutaneous Injection

SUMMARY:
This study is a clinical trial in patients with Parkinson's disease (PD), of a drug called exenatide, which is already licensed for the treatment of patients with type 2 diabetes. There have been several groups that have confirmed that exenatide has beneficial effects of nerve cells when tested in the laboratory, which raises the possibility that exenatide may slow down or stop the degeneration of PD. In an open label trial in patients with PD who self administered the drug for a period of 48 weeks, the investigators have previously shown that the drug is well tolerated and shows encouraging effects on the movement and non-movement aspects of the disease. A double blind placebo controlled trial involving 60 participants was then conducted which indicated that exenatide may be a "neuroprotective" drug, i.e. one that stops the nerve cells dying in PD. The next step is therefore to confirm this "neuroprotective" effect and to see whether this effect can be reproduced in a multi-centre setting including a larger number of participants. An important objective is to explore whether any positive effects remain static or increase when the treatment is continued over a 96 week period. In order to explore this, a randomised, double blind, parallel group, placebo controlled, Phase 3 trial of Exenatide is being undertaken (Exenatide-PD3).

DETAILED DESCRIPTION:
This study is a clinical trial in patients with Parkinson's disease (PD), of a drug called exenatide, which is already licensed for the treatment of patients with type 2 diabetes. There have been several groups that have confirmed that exenatide has beneficial effects of nerve cells when tested in the laboratory, which raises the possibility that exenatide may slow down or stop the degeneration of PD. In an open label trial in patients with PD who self administered the drug for a period of 48 weeks, investigators have previously shown that the drug is well tolerated and shows encouraging effects on the movement and non-movement aspects of the disease. A double blind placebo controlled trial involving 60 participants was then conducted which indicated that exenatide may be a "neuroprotective" drug, i.e. one that stops the nerve cells dying in PD. The next step is therefore to confirm this "neuroprotective" effect and to see whether this effect can be reproduced in a multi-centre setting including a larger number of participants. An important objective is to explore whether any positive effects remain static or increase when the treatment is continued over a 96 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease.
2. Hoehn and Yahr stage ≤2.5 in the ON medication state.
3. Between 25 and 80 years of age.
4. On dopaminergic treatment for at least 4 weeks before enrolment.
5. Ability to self-administer, or to arrange carer administration of trial medication.
6. Documented informed consent to participate.

Exclusion Criteria:

1. Diagnosis or suspicion of other cause for Parkinsonism.
2. Patients unable to attend the clinic visits in the practically defined OFF medication state.
3. Body mass index <18.5.
4. Known abnormality on CT or MRI brain imaging considered likely to compromise compliance with trial protocol.
5. Significant cognitive impairment defined by a score <21 on the Montreal Cognitive Assessment.
6. Concurrent severe depression defined by a score ≥16 on the Patient Health Questionnaire (PHQ-9).
7. Prior intra-cerebral surgical intervention for Parkinson's disease.
8. Previous participation in one of the following Parkinson's disease trials (Biogen SPARK trial, Prothena Pasadena trial, Sanofi Genzyme MOVES-PD trial, UDCA-PD UP Study or any other trial still considered to involve a potentially PD modifying agent).
9. Participation in another clinical trial of a device, drug or surgical treatment within the last 30 days
10. Previous exposure to exenatide.
11. Impaired renal function with creatinine clearance <50ml/min.
12. History of pancreatitis.
13. Type 1 or Type 2 diabetes mellitus.
14. Severe gastrointestinal disease (e.g. gastroparesis)
15. Hyperlipidaemia.
16. History or family history of medullary thyroid cancer (MTC).
17. Multiple endocrine neoplasia 2 (MEN2) syndrome.
18. Hypersensitivity to any of exenatide's excipients.
19. Females that are pregnant or breast feeding.
20. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire trial period and up to 3 months after the last dose of trial medication.
21. Participants who lack the capacity to give informed consent
22. Any medical or psychiatric condition or previous conventional/experimental treatment which in the investigator's opinion compromises the potential participant's ability to participate.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-02-24 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3 | 96 weeks
  Comparison of MDS-UPDRS part 3 motor sub-score in the practically defined OFF medication state at 96 weeks between participants according to treatment allocation. Min value- 0 Max Value- 108. Higher score indicative of worse outcome.

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale part 1,2, and 4 ON medication scores. | 96 weeks
  Questionnaire. Section I: 16 points; Section II: 52; Section IV: 23. Higher score indicative of worse outcome.
Timed Walk assessment ON and OFF medication | 96 weeks
  Assessment with research team
Montreal Cognitive Assessment | 96 weeks
  Questionnaire. Maximum Score= 30. Lower scores indicative of worse outcome.
Unified Dyskinesia Rating Scale (UDysRS) | 96 weeks
  Questionnaire. The UDysRS has four parts: I: Historical Disability (patient perceptions) of On-Dyskinesia impact (maximum 44 points); II: Historical Disability (patient perceptions) of Off-Dystonia impact (maximum 16 points); III: Objective Impairment (dyskinesia severity, anatomical distribution over seven body regions, and type (choreic or dystonic) based on four activities observed or video-recorded (28 points); IV: Objective Disability based on Part III activities (maximum 16 points). Higher scores= worse outcomes
Patient Health Questionnaire-9 (PHQ-9) | 96 weeks
  Questionnaire. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Max Score= 27. Higher Score= worse outcome
Parkinson's Disease 39 item Quality of life questionnaire | 96 weeks
  This questionnaire assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. The 39 item questionnaire offers a patient reported measure of health status and quality of life and is the most frequently used disease-specific health status measure. Higher score= worse outcome.
Non-Motor Symptoms Scale (NMSS) | 96 weeks
  Questionnaire. The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients at all stages of PD. Higher score indicative of worse outcome. NMSS total score is 0 to 360.
Levodopa Equivalent Dose | 96 weeks
  Assessment with Research Team
3 day Hauser diary of Parkinson's Disease State | 96 weeks
  Participant take Home questionnaire. (Time-On, Off, Non troublesome Dyskinesia, Troublesome dyskinesia, Asleep). Higher total scores indicate more severe motor signs of Parkinson's.
Safety and tolerability of exenatide as indicated by changes in pulse (bpm) | 96 weeks
  Vital Signs
Safety and tolerability of exenatide as indicated by changes in blood pressure (mmHg) | 96 weeks
  Vital Signs
Safety and tolerability of exenatide as indicated by changes in Body Mass Index (weight and height will be combined to report BMI in kg/m^2) | 96 weeks
  Vital Signs
Safety and tolerability of exenatide as indicated by changes in Red Blood Cell Count (10^12/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in White Blood Cell Count (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Haemoglobin (g/dL) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Haematocrit (%) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Platelets (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Neutrophils (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Eosinophils (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Basophils (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Lymphocytes (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Monocytes (10^9/L) | 96 weeks
  Full Blood Count
Safety and tolerability of exenatide as indicated by changes in Prothrombin Time (secs) | 96 weeks
  Blood Tests (Coagulation)
Safety and tolerability of exenatide as indicated by changes in International Normalized Ratio (Calculated from Prothrombin Time) | 96 weeks
  Blood Tests (Coagulation)
Safety and tolerability of exenatide as indicated by changes in Activated Partial Thromboplastin Time (secs) | 96 weeks
  Blood Tests (Coagulation)
Safety and tolerability of exenatide as indicated by changes in Thrombin Time (secs) | 96 weeks
  Blood Tests (Coagulation)
Safety and tolerability of exenatide as indicated by changes in Fibrinogen (g/L) | 96 weeks
  Blood Tests (Coagulation)
Safety and tolerability of exenatide as indicated by changes in Glycated Haemoglobin (% of Haemoglobin) | 96 weeks
  Blood Tests (Blood Sugar Levels / Diabetes Testing)
Safety and tolerability of exenatide as indicated by changes in Sodium (mmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Potassium (mmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Urea (mmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Creatinine (µmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Creatinine Clearance (ml/min) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Total Bilirubin (µmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Alkaline phosphatase (IU/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Alanine transaminase (IU/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Aspartate Aminotransferase (IU/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Serum Amylase (U/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Thyroid Stimulating Hormone (mIU/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Thyroxin (T4) (pmol/L) | 96 weeks
  Biochemistry
Safety and tolerability of exenatide as indicated by changes in Triglycerides (mg/dL) | 96 weeks
  Biochemistry (Fasting)
Safety and tolerability of exenatide as indicated by changes in Cholesterol (mg/dL) | 96 weeks
  Biochemistry (Fasting)
Safety and tolerability of exenatide as indicated by changes in Glucose (mmol/L) | 96 weeks
  Biochemistry (Fasting)
Safety and tolerability of exenatide as indicated by changes in Insulin (IU/L) | 96 weeks
  Biochemistry (Fasting)
Safety and tolerability of exenatide as indicated by the occurrence / severity of Adverse Events | 96 weeks
  Ongoing Safety Reporting

CONTACTS AND LOCATIONS:
Overall Officials: Tom Foltynie, Principal Investigator — University College London Comprehensive Clinical Trials Unit
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vijiaratnam N, Girges C, Auld G, McComish R, King A, Skene SS, Hibbert S, Wong A, Melander S, Gibson R, Matthews H, Dickson J, Carroll C, Patrick A, Inches J, Silverdale M, Blackledge B, Whiston J, Hu M, Welch J, Duncan G, Power K, Gallen S, Kerr J, Chaudhuri KR, Batzu L, Rota S, Jabbari E, Morris H, Limousin P, Greig N, Li Y, Libri V, Gandhi S, Athauda D, Chowdhury K, Foltynie T. Exenatide once a week versus placebo as a potential disease-modifying treatment for people with Parkinson's disease in the UK: a phase 3, multicentre, double-blind, parallel-group, randomised, placebo-controlled trial. Lancet. 2025 Feb 22;405(10479):627-636. doi: 10.1016/S0140-6736(24)02808-3. Epub 2025 Feb 4. PMID 39919773
- [Derived] Vijiaratnam N, Girges C, Auld G, Chau M, Maclagan K, King A, Skene S, Chowdhury K, Hibbert S, Morris H, Limousin P, Athauda D, Carroll CB, Hu MT, Silverdale M, Duncan GW, Chaudhuri R, Lo C, Del Din S, Yarnall AJ, Rochester L, Gibson R, Dickson J, Hunter R, Libri V, Foltynie T. Exenatide once weekly over 2 years as a potential disease-modifying treatment for Parkinson's disease: protocol for a multicentre, randomised, double blind, parallel group, placebo controlled, phase 3 trial: The 'Exenatide-PD3' study. BMJ Open. 2021 May 28;11(5):e047993. doi: 10.1136/bmjopen-2020-047993. PMID 34049922
- See also: Sponsor Trial web link — https://www.ucl.ac.uk/comprehensive-clinical-trials-unit/research-projects/2021/jan/exenatide-parkinsons-disease